CLINICAL TRIAL: NCT06034210
Title: The Effectiveness of Customised 3D-printed Insoles on Perceived Pain, Comfort, and Completion Time Among Frequent Park Runners: A Pragmatic Randomised Controlled Trial (The ZOLES Trial)
Brief Title: Effectiveness of Customised 3D-printed Insoles in Reducing Pain Among Frequent Park Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's University, Twickenham (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Aalborg University (Other); Zoles ApS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZolesRCT
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZOLES insoles (Experimental): Participants allocated to the intervention group will receive customised 3D-printed insoles (Zoles ApS, Espergærde, DK-3060, Denmark) to mitigate running-related pain and discomfort. Being a pragmatic trial, all participants are permitted to continue or initiate any usual care of their choice.
  Interventions: Device: Customised 3D-printed insoles
- Do-as-usual (No Intervention): Participants allocated to the control group are a "do-as-usual" comparator. This implies, that the participants can treat and prevent running-related pain and discomfort in any way they wish, except using the Zoles 3D-printed insoles.

INTERVENTIONS:
Device: Customised 3D-printed insoles — Based on measurements from the 3D scanning procedure, and factoring in individual data such as age, weight, and activity preferences, custom insoles are designed using the ZOLA software. The insoles are then 3D-printed by Zoles ApS in Espergærde (Denmark), using BCN3D printers (Barcelona, Spain) and a TPU (Thermoplastic Polyurethane) filament material from Recreus (Alicante, Spain). The printed insoles are tailored for optimal support, performance, and comfort, with varying densities for areas like the arch and heel. They are finished with an OnSteam® microfiber cover for added durability and comfort. The insoles are intended for regular insertion into participants' shoes to align with their unique biomechanical needs. (Information translated and adapted from: https://www.zoles.eu/da/processen-bag-saalerne/)
  Other Names: Zoles insoles
  Arms: ZOLES insoles

SUMMARY:
This study evaluates the effectiveness of the Zoles customised 3D-printed insoles to mitigate running-related pain among frequent recreational runners who participate in regular Park Run activities. All participants will have their feet scanned, after which half of the participants will be provided with customised 3D-printed insoles, while the other half will receive no intervention.

DETAILED DESCRIPTION:
The ZOLES trial is a pragmatic, outcome assessor blinded, randomised, controlled, superiority trial, with a two-group parallel design. Frequent recreational runners who participate in regular Park Run activities will undergo a foot scanning after which they will be randomised in a 1:1 allocation ratio to either receive a customised 3D-printed insole (Zoles ApS, Espergærde, DK-3060, Denmark), or to be in a "do-as-usual" control group. It is expected that the allocated intervention group participants will have received their customised insoles around two weeks after baseline during the follow-up period (one week to manufacture, one week to distribute). The primary endpoint is change in running-related pain 10 weeks after baseline (∼8 weeks after receiving allocated intervention).

A full trial protocol, based on the "SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials" and the "PREPARE Trial guide", will be published and made publicly available. The trial report will follow the "REPORT guide", and thus adhere to the CONSORT guidelines for reporting parallel group randomised trials, using the CONSORT extension for pragmatic trials, as well as the updated CONSORT-Outcomes 2022 extension. The TIDieR template is used to describe the intervention to aid future replication.

The central aim of this study is to establish the effectiveness of the Zoles customised 3D-printed insoles in alleviating running-related pain among frequent recreational runners participating in regular Park Run activities when compared against a "do-as-usual" control group. This clinical effectiveness will be reported in the main trial paper, which also includes the following key secondary outcomes: Global Rating of Change (GRoC) in overall daily pain and discomfort, Running-related foot/footwear comfort, 5-k (Park Run) completion time, running-related injury incidence rate, Time-loss from running, running exposure in miles and time, adherence to the intervention during daily- and running activities, and adverse events from using the Zoles insoles. Missing values will be imputed using multiple imputations by chained equations based on the following variables: All previous scores within the relevant outcome category, Age, Sex, Group Allocation, and enrolment (Park Run) location.

A total of 200 participants are anticipated to be enrolled, resulting in a minimum of 100 participants in each arm. The enrolment concludes once at least 100 participants have been allocated to each arm. Being a pragmatic trial, the eligibility criteria are loosely defined such that participants should simply be regular runners engaged in frequent Park Run activities, at a minimum 35 years of age. The participants will undergo balanced block randomization (1:1 allocation ratio), ensuring stratification for sex and enrolment location. The trial will include prospective weekly data collection using e-mail-distributed surveys via REDCap (Vanderbilt University, Nashville, TN, USA) throughout the 10-week follow-up period. After the conclusion of the initial 10-week trial phase, the control group will also be provided with their customised 3D-printed insoles. This will not be weekly monitored, however, following an additional 8-week period with the insoles, this group will then complete the follow-up questionnaire again, to ascertain whether similar benefits or deterioration from the insoles in a manner consistent with the original experimental group are experienced. At the conclusion of the trial, and as part of a post-market surveillance approach, all participants, both from the original experimental and control groups (who by this point have received the intervention), will be administered a final questionnaire after a 1-year period to evaluate the long-term effects and durability of the benefits associated with the customised 3D-printed insoles.

The primary outcome; change in running-related pain from baseline to follow-up, will be calculated using negative binomial regression, adjusting for values reported at baseline. Both the Global Rating of Change (GRoC) in overall daily pain and discomfort, and Running-related foot/footwear comfort will be calculated similarly. Injury incidence rate ratios will be estimated per 1000 hours of running exposure using Poisson regression. Mean time-loss from running will be calculated using negative binomial regression. Adherence to the intervention will be descriptively analysed and presented, and adverse event due to the Zoles insoles will be presented in type and frequency. Every analysis in the main trial report will abide by the intention to treat principle, which means including all participants in the analyses, regardless of intervention adherence-signifying that participants will be analyzed based on initial randomization. In the primary trial report, all collected outcomes will be listed, and it will also be stated that the below-mentioned 'other pre-specified outcomes' will be reported in a subsequent secondary analysis publication with a clear reference to the primary trial registration.

The subsequent secondary analysis publication will hold the label "secondary and long-term follow-up analysis from a pragmatic randomized controlled trial" in the title. The aims of this secondary subgroup analysis study are two-fold: First, it is to investigate the immediate therapeutic effect of Zoles insoles, focusing only on participants with clinically relevant baseline pain levels (11-NRS ≥ 3). Secondly, this will include our long-term post-market analysis to evaluate the long-term effects and durability of the benefits associated with the customised 3D-printed insoles one year post-intervention. In the secondary subgroup analysis, the following outcomes will be reported: Percentage of participants achieving a change of at least MCID (11-NRS ≥ 2) in running-related pain, Time until change in running-related Pain of at least MCID, Change among participants with clinically relevant running-related pain at baseline, Pre-trial expectations to the therapeutic effect of using the Zoles insoles, and Post-trial experiences on the therapeutic effect of using the Zoles insoles. Incorporating the expectations and post-intervention experiences as covariates, regression models will be constructed to understand the potential influence of these factors on the efficacy of the Zoles insoles intervention within this specific subgroup of participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 35 years old at commencement of trial
* Participant can read, speak and understand English
* Participant can receive e-mails and complete online questionnaires
* Participant is a frequent runner who participate in regular Park Runs
* Participant is capable of running at commencement of trial

Exclusion Criteria:

* Individuals with severe foot deformities
* Individuals with uncontrolled diabetes with foot complications, or other conditions that might interfere with their ability to safely use the insoles and participate in running activities

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Running-related Pain | 10 weeks
  Change in running-related pain from baseline to follow-up during the trial period. Pain is scored on a numeric rating scale from 0 - 10 (0 = No pain at all, 10 = Extremely painful; Salaffi et al., 2004)

SECONDARY OUTCOMES:
Global Rating of Change (GRoC) in overall daily pain and discomfort | 10 weeks
  Participants' self-perceived change in overall daily pain and discomfort in relation to when they were enrolled in the study. Participants rate their perceived improvement or deterioration on a 7-point scale ranging from -3 = "much worse" to 3 = "much better" (Bobos et al., 2019)
Running-related foot/footwear comfort | 10 weeks
  Change in running-related foot/footwear comfort from baseline to follow-up during the trial period. Comfort is scored on a numeric rating scale from 0 - 10 (0 = Extremely uncomfortable, 10 = Extremely comfortable; Menz & Bonnano, 2021)
5k-completion time | 10 weeks
  Time in minutes taken to complete the weekly 5 km Park Run at their chosen Park Run location
Running-related injuries | 10 weeks
  Rate of running-related injuries sustained during the trial period. The incidence rate is defined as the number of injuries per 1000 hours of running exposure
Time-loss | 10 weeks
  Time lost from running in number of days due to running-related pain, discomfort, or injury
Weekly Milage | 10 weeks
  Weekly distance covered from running activities during the trial period
Weekly running exposure | 10 weeks
  Weekly exposure to running activities in hours and minutes during the trial period
Adherence to intervention, ADL% | 10 weeks
  Relative use of the Zoles insoles during all sitting/standing/walking/driving activities
Adherence to intervention, RUN% | 10 weeks
  Relative use of the Zoles insoles during all running activities
Adverse events from using Zoles insoles | 52 weeks
  Adverse events will be reported as type and number of events. The included participants will be encouraged to report any adverse events related to the use of Zoles via the trial hotline

OTHER OUTCOMES:
Participants achieving MCID reduction in pain | 10 weeks
  Percentage of participants achieving a change in running-related pain of at least the size of MCID (NRS ≥ 2, Salaffi et al., 2004) during the trial intervention period
Time until MCID reduction in pain | 10 weeks
  Time until change in running-related Pain of at least MCID. Time in weeks until a change in running-related pain of at least the size of MCID (NRS ≥ 2, Salaffi et al., 2004) during the trial intervention period, for participants with clinically relevant levels of pre-existing pain (NRS ≥ 3, Rathleff et al., 2019) during running-related activities
Change among participants with high baseline pain | 10 weeks
  Change in running-related pain from baseline to follow-up during the trial period for participants with clinically relevant pre-existing pain levels of NRS ≥ 3 (Rathleff et al., 2019) during running activities. Pain is scored on a numeric rating scale from 0 - 10 (0 = No pain at all, 10 = Extremely painful)
Pre-trial intervention expectations | 52 weeks
  Pre-trial expectations to the therapeutic effect of using the Zoles insoles. The participants' expected effects of the insole intervention on running-related pain, 5-k completion time, and foot/footwear comfort are reported at baseline using 5-point Likert scales ranging from "significantly worsen" to "significantly improve"
Post-trial intervention experiences | 52 weeks
  Post-trial experiences on the therapeutic effect of using the Zoles insoles. Post-intervention period, the participants are asked on whether the intervention met, exceeded, or did not meet their expectations using a 5-point Likert scale ranging from "Fell well short of expectations" to "greatly exceeded expectations"
Post-market surveillance | 52 weeks
  Post-market surveillance including the primary outcome and all key secondary outcomes. All participants, both intervention and control groups will be administered a final questionnaire after a 1-year period to evaluate the long-term effects and durability of the benefits associated with the customised 3D-printed insoles

CONTACTS AND LOCATIONS:
Overall Officials: Filip Gertz Lysdal, MSc, PhD, Study Director — Faculty of Sport, Technology and Health Sciences, St Mary's University, United Kingdom; Suleyman Ibrahim, MEd, Principal Investigator — Faculty of Sport, Technology and Health Sciences, St Mary's University, United Kingdom; Chris Djurtoft, PT, MSc, Study Chair — Department of Clinical Medicine, Aalborg University, Denmark; Rik Mellor, MSc, Study Chair — Faculty of Sport, Technology and Health Sciences, St Mary's University, United Kingdom; Kristian Thorborg, PT, MSc, PhD, Study Chair — Sports Orthopaedic Research Center-Copenhagen (SORC-C), Department of Orthopaedic Surgery, Copenhagen University Hospital, Amager-Hvidovre, Denmark
Locations (1):
- St Mary's University, Faculty of Sport, Technology and Health Sciences, Twickenham, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim S, Djurtoft C, Mellor R, Thorborg K, Lysdal FG. The effectiveness of customised 3D-printed insoles on perceived pain, comfort, and completion time among frequent Park Runners: Study protocol for a pragmatic randomised controlled trial (The ZOLES RCT). Foot (Edinb). 2024 Mar;58:102068. doi: 10.1016/j.foot.2024.102068. Epub 2024 Feb 6. PMID 38350194

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT06034210/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT06034210/ICF_001.pdf